CLINICAL TRIAL: NCT04360967
Title: Neurodevelopment, Growth, and Metabolic Syndrome Biomarkers in Term Small-for-gestational-age Infants Fed Standard or Nutrient-enriched Formula
Brief Title: SURF, Neurodevelopment, Growth Study in SGA Infants
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision stopped in June 2017
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 14.11.INF
Record Dates: First submitted 2017-01-10; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Infant, Small for Gestational Age

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Randomized Standard Formula-fed (Experimental): Product will be given to the formula-fed groups during the intervention phase of the study (enrollment to age 6 months).
  Interventions: Other: Standard Formula
- Randomized Nutrient-enriched formula-fed (Experimental): Product will be given to the formula-fed groups during the intervention phase of the study (enrollment to age 6 months).
  Interventions: Other: Nutrient-enriched Formula
- Non-randomized HM-fed (No Intervention): Infants in HM-fed group will be fed through 6 months of age, along with micronutrient supplementation per routine clinical practice.
- Non-Randomized HM-fed (No Intervention): Infants in HM-fed group will be fed through 6 months of age, along with micronutrient supplementation per routine clinical practice.

INTERVENTIONS:
Other: Standard Formula — Standard Formula
  Arms: Randomized Standard Formula-fed
Other: Nutrient-enriched Formula — Nutrient-enriched Formula
  Arms: Randomized Nutrient-enriched formula-fed

SUMMARY:
The purpose of this study is to determine whether term SGA infants who are fed a nutrient-enriched pre-term formula will have a higher cognitive score, a more appropriate length-for-age Z-score (leading to a lower prevalence of Stunting) but higher blood pressure at 2 years of age compared to term SGA infants who are fed on a regular starter formula.

DETAILED DESCRIPTION:
This is multi-sites, interventional, double-blinded, randomized, 2-arm parallel-group clinical trial. Two HM fed groups will be included as comparator group.

The primary objectives are:

1. To evaluate neurodevelopment at 2 years of age in term small-for-gestational age (SGA) infants fed standard formula or nutrient-enriched formula from 1 to 6 months of age and compare to each human milk (HM)-fed group.
2. To evaluate length-for-age Z-score at 2 years of age in term SGA infants fed standard formula or nutrient-enriched formula from 1 to 6 months of age and compare to each HM-fed group.
3. To evaluate systolic blood pressure at 2 years of age in term SGA infants fed standard formula or nutrient-enriched formula from 1 to 6 months of age and compare to each HM-fed group.

ELIGIBILITY:
Inclusion Criteria:

1. Having obtained his/her parents' (or his/her legally accepted representative's LAR's]) written informed consent and having evidence of a personally signed and dated informed consent document indicating that the infant's parents/LAR have been informed of pertinent aspects of the study.
2. For infants in formula fed groups only: infants who require formula feeding due to lactation failure after minimum 2 rounds of breastfeeding counselling.
3. Birth Weight < 10th percentile at term using the 2013 INTERGROWTH-21st Growth Charts for girls and boys.
4. Full term birth (gestational age ≥ 37 weeks and ≤ 41 weeks + 6 days), with gestational age estimated using fetal anthropometry by ultrasonography in early 1st trimester of pregnancy or calculated using the first day of the last menstrual period + 40 weeks if fetal anthropometry data for term calculation is not available or was collected after the 1st trimester.
5. Age <45 days at time of enrollment
6. For infants in the HM-fed AGA comparator group only: born to mothers with pre-pregnancy body mass index (BMI) ≥ 18.5 and <25kg/m2

Exclusion Criteria:

1. mothers with Type-1 Diabetes
2. mothers who smoked >10 cigarettes per day during pregnancy.
3. mothers who used Illicit drugs (e.g. marijuana, cocaine, amphetamines, or heroin) or alcohol (>3 alcoholic beverages per week) during pregnancy
4. Suspected or documented systemic or congenital infections (e.g Human Immunodeficiency virus, cytomegalovirus)
5. Genetic or any other type of congenital malformations, metabolic, cardiovascular, gastrointestinal, pancreatic or hepatic diseases or medical conditions that could compromise growth and/or food intake.
6. Fit to be discharged from neonatal intensive care unit (NICU) in > 5 consecutive days with the exception of infants in the NICU due to jaundice only.
7. Known or suspected intolerance/ allergy to milk protein or any ingredient in the study formulas
8. For infants in the HM-fed groups only: infants who are consuming fortified human milk or formula.
9. Participation in any other interventional clinical trial during the 14 days prior to enrollment.
10. Infants or infant's family who in the investigator's judgement cannot be expected to comply with the protocol or study procedures.

Ages: 1 Day to 44 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2017-03-31 (Estimated); Primary Completion 2017-06-02 (Estimated); Study Completion 2017-06-02 (Estimated)

PRIMARY OUTCOMES:
Evaluation of neurodevelopment | at the baseline (2 years of age)
  Assessed using Bayley Scales of Infant and Toddler Development® - Third Edition - (To compare with the standard Bayley scores).
Evaluation of length-for-age Z-score | Evaluated once at 2 years of age
  Using the WHO growth chart
Systolic Blood pressure | at baseline (2 years of age)
  Systolic and diastolic blood pressure measurement from 1 to 6 months of age

SECONDARY OUTCOMES:
Evaluation of insulin sensitivity | at Baseline ( 2 years of age).
  HOMA-IR (Homeostatic Model Assessment - Insulin Resistance) calculated from Basal (Fasting) plasma glucose and insulin concentrations.
Evaluation of insulin sensitivity | at last visit ( 5 years of age).
  HOMA-IR (Homeostatic Model Assessment - Insulin Resistance) calculated from Basal (Fasting) plasma glucose and insulin concentrations.
Neurodevelopment | At last visit ( 5 years of age)
  Assessed using Wechsler Preschool and Primary Scale of Intelligence™ - Fourth Edition (WPPSI-IV) - (to compare the scores against the standard scores).
Safety (Adverse Event reporting) | From 1 to 6 months of age & 6 months to 5 years of age.
  Assessed by Type, incidence, severity, seriousness and relationship to study formulas of AEs (including Infection) among the study subjects.
Growth (Length) | At 2 years of age
  Evaluation of length-for-age in each formula-fed group by Percentages of study population with length-for-age Z-score less than 2.5th, 5th and 10th Percentile on the WHO reference curve(<2.5th percentile indicating prevalence of stunting).
Growth (Weight) | At 2 years of age
  Evaluation of weight-for-age in each formula-fed group by Percentages of study population with length-for-age Z-score less than 2.5th, 5th and 10th Percentile on the WHO reference curve(<2.5th percentile indicating prevalence of stunting).
Growth (Head circumference) | At 2 years of age
  Evaluation of head circumference-for-age in each formula-fed group by Percentages of study population with length-for-age Z-score less than 2.5th, 5th and 10th Percentile on the WHO reference curve(<2.5th percentile indicating prevalence of stunting).
Growth (Z-Scores) | At 2 years of age
  Evaluation of weight-for-length Z-scores in each formula-fed group by Percentages of study population with length-for-age Z-score less than 2.5th, 5th and 10th Percentile on the WHO reference curve(<2.5th percentile indicating prevalence of stunting).
Evaluation of serum markers of bone metabolism | At visit 1 (<44 days)
  Assessed by Incidence of abnormal serum (Calcium, phosphorus, Alkaline phosphatase).
Evaluation of serum markers of bone metabolism | At visit 4 (6 months)
  Assessed by Incidence of abnormal serum (Calcium, phosphorus, Alkaline phosphatase).
Evaluation of urinary markers of bone metabolism | At visit 1 (<44 days)
  Assessed by Incidence of urine biochemistries (calcium, phosphorous).
Evaluation of urinary markers of bone metabolism | At visit 4 (6 months)
  Assessed by Incidence of urine biochemistries (calcium, phosphorous).
Body fat mass (%) | evaluated until 5 years of age.
  Assessed by Deterium dilution

IPD SHARING:
Plan to Share IPD: Undecided